CLINICAL TRIAL: NCT04914637
Title: The Effect of Dry Needling on the Treatment Outcomes of Interlaminar Epidural Steroid Injection in Patients With Chronic Neck Pain Due to Cervical Disc Herniation.
Brief Title: Does Dry Needling Affect Treatment Outcomes of Interlaminar Epidural Steroid Injection in Cervical Disc Herniation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2020.692
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pain, Myofacial; Pain, Neck; Pain, Chronic
Keywords: myofascial trigger point pain; disc, herniated; epidural injections
MeSH Terms: conditions — Facial Pain; Neck Pain; Chronic Pain; Myofascial Pain Syndromes; Intervertebral Disc Displacement | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interlaminar epidural steroid injection plus dry needling (Active Comparator): Fluoroscopy-guided cervical interlaminar epidural steroid injection will be administered to patients with chronic neck pain due to cervical disc herniation. Also, dry needling will be applied to the active trigger points for the patients in this group.
  Interlaminar epidural steroid injection will be applied at week 0, while dry needling will be applied in 3 sessions per week (week 0, week 1, week 2). The first session of the dry needling will be in the same day with interlaminar epidural steroid injection.
  Interventions: Procedure: Cervical interlaminar epidural steroid injection; Procedure: Dry needling
- interlaminar epidural steroid injection plus sham dry needling (Sham Comparator): Fluoroscopy-guided cervical interlaminar epidural steroid injection will be administered same as the arm titled "interlaminar epidural steroid injection plus dry needling". The only difference in the interventions in this arm is that dry needling is applied without penetrating the skin. The blunt tip of the needle will be used in sham intervention.
  Interlaminar epidural steroid injection will be applied at week 0, while sham dry needling will be applied in 3 sessions per week (week 0, week 1, week 2)
  Interventions: Procedure: Cervical interlaminar epidural steroid injection; Procedure: Sham dry needling
- interlaminar epidural steroid injection only (Other): Only interlaminar epidural steroid injection will be administered to patients in this arm with the same method as in the other arms (one session, week 0). No dry needling or sham dry needling will be used.
  Interventions: Procedure: Cervical interlaminar epidural steroid injection

INTERVENTIONS:
Procedure: Cervical interlaminar epidural steroid injection — Fluoroscopy-guided cervical interlaminar epidural steroid injection will be administered to patients with chronic neck pain due to cervical disc herniation. The injection area is cleaned 3 times with an antiseptic solution and covered with a sterile cloth. Local anesthesia with 2 cc 3% prilocaine will be applied to the skin and subcutaneous tissues in the area of interest. Under fluoroscopy guidance, the needle is advanced into the C7-T1 intervertebral disc level. With the help of the loss of resistance technique, it is understood that the needle is in the epidural space, and second control is provided by administering contrast material. After the confirmation of needle place is done, a mixture of 12 mg dexamethasone, 1 cc 2% lidocaine, 1 cc saline is injected. The patient is taken to the rest room after the procedure and followed up for any complications.
Procedure: Dry needling — Dry needling will be applied to the active trigger points for the patients in this group. After cleaning the area of interest with an antiseptic solution, dry needling will be applied with the fast-in/fast-out technique for the active trigger point. During needle maneuvers, local contractions (local twitch response-LTR) are obtained and rapid needle movements are continued until the contractions end. Afterwards, the needle is removed and compression is applied to ensure hemostasis in the relevant area.
  Arms: interlaminar epidural steroid injection plus dry needling
Procedure: Sham dry needling — Although the method of intervention is like dry needling, the only difference is that the blunt end of the needle is used and it does not penetrate the skin.
  Arms: interlaminar epidural steroid injection plus sham dry needling

SUMMARY:
Chronic neck pain is among the most frequently seen chronic painful conditions. As an important cause of disability, chronic neck pain is a musculoskeletal disorder that negatively affects quality of life. Cervical disc herniation is one of the leading causes of chronic neck pain and conservative methods such as exercise and pain medications are used first in the treatment. In patients unresponsive to conservative treatment, epidural steroid injection is successfully and frequently used treatment option. Epidural steroid injection in the cervical region can be applied with two approaches: interlaminar or transforaminal.

Myofascial trigger point characterized by intramuscular taut band and hypersensitive spots is a condition in which central and peripheral sensitization play a role in the pathophysiology. There are underlying myofascial trigger points in many etiologies that cause chronic neck pain. Trigger points can increase the severity of pain and in some cases they can be the main factor in the etiology of pain. Therefore, the presence of myofascial trigger points should be investigated, even if another cause is detected in chronic neck pain. Dry needling is an easily applicable and effective treatment option in myofascial trigger point.

Although it is well known that myofascial trigger points frequently accompany cervical disc herniation, their effect on treatment outcomes has not been investigated. In this study, we aimed to investigate the effect of dry needling for trigger points on the treatment results of interlaminar epidural steroid injection in patients diagnosed with cervical disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Chronic neck pain due to cervical disc herniation for at least 3 months and being unresponsive to conservative treatment
* Presence of at least one active myofascial trigger point on physical examination of cervical paraspinal muscles, scapulothoracic muscles and extremity muscles.

Exclusion Criteria:

* Previous surgical/interventional procedure for the cervical region
* Previous application of dry needling/acupuncture to any part of the body
* Presence of other musculoskeletal disorders (such as lateral epicondylitis, tendinitis, entrapment neuropathy) that may cause diagnostic confusion in terms of pain pattern and localization
* Signs of trauma, fracture, malignancy, or active infection
* Rheumatological (RA, AS, etc.), endocrinological (such as osteoporosis, Paget's disease) or another systemic disease that may change the anatomical or physiological structure of the relevant regions
* Presence of coagulopathy
* History of whiplash injury, cervical spinal stenosis, cervical spondylosis
* Have a diagnosis of fibromyalgia
* Being pregnant and breastfeeding
* Presence of mental deterioration or psychiatric/neurological disease that can affect flow of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Change of pain severity from baseline to each checkpoints | from pre-interventional time to post-interventional 1st hour, 3rd week, 3rd month
  Pain severity will be assessed with Numeric Rating Scale (NRS). The patient scores his/her pain between 0-10. Higher score indicates more severe pain
Change of the number of active trigger points from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  The number of active trigger points will be determined by clinical examination. The trigger point will be defined as "active" if it causes spontaneous pain or pain occured during the examination is familiar to the patient.

SECONDARY OUTCOMES:
Change of depression severity from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  Severity of depression will be assessed with Beck Depression Inventory (BDI). BDI scoring ranges from 0 to 63, with a high score indicating an increased severity of depression.
Change of the number of the patients with neuropathic pain from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  The number of patients with neuropathic pain will be assessed with Douleur Neuropathique 4 Questions (DN4). Scores ≥ 4/10 indicate presence of neuropathic pain.
Change of the number of the patients with central sensitization from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  The number of patients with central sensitization will be assessed with The number of patients with neuropathic pain will be assessed with Central Sensitisation Inventory (CSI). The CSI is composed of two parts: Part A and part B. Only Part A is scored and a score of more than 40 indicates the presence of central sensitisation.
Change of the measurement of quality of life from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  The measurement of quality of life will be assessed with Short Form-12 Survey (SF-12). Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). A high score indicates better quality of life.
Change of the measurement of disability related with chronic neck pain from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  The measurement of disability will be assessed with Neck Disability Index (NDI). The NDI can be scored as a raw score (0-50) or doubled and expressed as a percent (0%-100%). A higher score indicates more activity limitation.
Change of the measurement of sleep quality from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  The measurement of sleep quality will be assessed with Pittsburgh Sleep Quality Index (PSQI). 7 components are evaluated and each component is scored between 0-3; the total score is between 0-21. Higher total score indicates poor sleep quality.
Change of the pain sensitivity of active trigger points from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  The measurement of pain sensitivity will be done by using manual algometer. Measurement will be made from active trigger points and the average of 3 measurements will be taken. The higher score indicates more resistance to pain.

CONTACTS AND LOCATIONS:
Overall Officials: Osman Hakan Gunduz, MD, Principal Investigator — Marmara University
Locations (1):
- Marmara University Pendik Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yolcu G, Toprak CS, Sencan S, Gunduz OH. Dry Needling Plus Cervical Interlaminar Epidural Steroid Injections: Do We Have More Favorable Results in Cervical Disc Herniation? A Randomized Sham-Controlled Clinical Study. Am J Phys Med Rehabil. 2024 Dec 1;103(12):1081-1087. doi: 10.1097/PHM.0000000000002509. PMID 39671525